CLINICAL TRIAL: NCT04064671
Title: ZEPHYR: A Prospective Study Evaluating Surgical Outcome After Implantation of the Zephyr ZSI 475 FTM Inflatable Penile Implant in the Neophallus After Female-to-male Sex Reassignment Surgery
Brief Title: ZEPHYR: A Study Evaluating Surgical Outcome After Implantation of the Zephyr ZSI 475 FTM Inflatable Penile Implant in the Neophallus After Female-to-male Sex Reassignment Surgery
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/0025 (BC-4486)
Record Dates: First submitted 2019-08-07; First posted 2019-08-22 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Erectile Dysfunction; Gender Dysphoria
Keywords: female-to-male; transgender; transsexual; Zephyr; erectile device; erectile implant; neophallus; phalloplasty; gender reassignment surgery; sex reassignment surgery
MeSH Terms: conditions — Erectile Dysfunction; Gender Dysphoria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Implantation of the Zephyr ZSI 475 FTM erectile implant — Until recently, all penile implants were manufactured for erectile dysfunction in biological males and thus presumed the presence of two corpora cavernosa. In 2016 however, the Swiss company, Zephyr Surgical Implants (ZSI), created a 3-piece inflatable erectile device specifically for female-to-male transsexuals: the Zephyr ZSI 475 FTM. This prosthesis has a realistic gland shape, only one cylinder, and a specific anchorage device made of titanium and silicone to anchor the system to the pubic bone of the patient. These specific features could potentially address the aforementioned issues with implanting erectile devices in the neophallus and hopefully lead to better surgical outcomes in these particular patients.

SUMMARY:
This study will look into the surgical outcome after implantation of the Zephyr ZSI 475 FTM in the neophallus.

DETAILED DESCRIPTION:
Obtaining erectile function after phalloplasty in female-to-male transsexuals remains a challenging issue and requires the implantation of a device. For biological males, several erectile implants exist and widespread research has demonstrated the successful outcome of these devices. However, substantial differences exist between a native penis and a neophallus and explain the poorer outcome of these devices in female-to-male transsexuals.

In 2018, Falcone et al. published the largest retrospective series on this subject so far and reported that after a mean follow-up of 20 months, only 58% of their patients still had their original implant in place. The main obstacle in these female-to-male transsexuals is represented by the lack of corpora cavernosa in the neophallus which leads to difficult anchorage of the prosthesis, little stability of the prosthesis and a higher risk of cylinder erosion.

Until recently, all penile implants were manufactured for erectile dysfunction in biological males and thus presumed the presence of two corpora cavernosa. In 2016 however, the Swiss company, Zephyr Surgical Implants (ZSI), created a 3-piece inflatable erectile device specifically for female-to-male transsexuals: the Zephyr ZSI 475 FTM. This prosthesis has a realistic gland shape, only one cylinder, and a specific anchorage device made of titanium and silicone to anchor the system to the pubic bone of the patient. These specific features could potentially address the aforementioned issues with implanting erectile devices in the neophallus and hopefully lead to better surgical outcomes in these particular patients.

So far, no literature regarding surgical or functional outcome of the Zephyr ZSI 475 FTM exists. The aim of this study is to prospectively collect data of all female-to-male transsexuals that are treated with the implantation of this device at Ghent University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed written informed consent according to the rules of Good Clinical Practice (Declaration of Helsinki) and national regulations.
* Age ≥ 18 years.
* Female-to-male transsexual patient.
* Implantation of Zephyr ZSI 475 FTM erectile device.

Exclusion Criteria:

* Absence of signed written informed consent.
* Age < 18 years.
* Biological males.
* Patients opting for penile implants other than the Zephyr ZSI 475 FTM.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — female-to-male transgenders after phalloplasty
Study Population: All female-to-male transsexual patients asking for the implantation of an erectile device are carefully counseled and during their visit, all available devices are discussed with their inherent benefits and drawbacks. If the patient independently chooses for the Zephyr ZSI 475 FTM erectile device, and if this patient meets the aforementioned inclusion criteria, he will be included in this study after voluntarily signing the written informed consent form.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-09-19 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Explantation-free survival | From date of surgery until the date of explantation or date of death from any cause, whichever came first, assessed up to 120 months postoperatively (assessment at 3 months postoperatively, 1 year postoperatively and then yearly)
  Interval between implantation date and explantation date (if explanted)

SECONDARY OUTCOMES:
Complication rate after implantation of this device | 90 days after implantation
  The Clavien-Dindo system (<90d) to report surgical complications will be used
Type of complications | From date of surgery until the date of explantation or date of death from any cause, whichever came first, assessed up to 120 months postoperatively (assessment at 3 months postoperatively, 1 year postoperatively and then yearly)
  Complications that will be assessed, involve:
  * Urinary tract infection (yes or no)
  * Hematuria (yes or no)
  * Wound infection (yes or no)
  * Wound dehiscence (yes or no)
  * Abscess formation (yes or no)
  * Fistula formation (yes or no)
  * Protrusion of the device (yes or no)
  * Malfunction of the device (yes or no)
  * migration of the device (yes or no)
  * Infection of the device (yes or no)

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Verla, Study Director — Dept. of Urology, Ghent University Hospital; Piet Hoebeke, Principal Investigator — Dept. of Urology, Ghent University Hospital
Locations (1):
- Department of Urology, Ghent University Hospital, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No